CLINICAL TRIAL: NCT04796363
Title: Ultrasound Guided Erector Spinae Plane Block in Breast Cancer Surgery: Analgesia, Spread and Immunomodulation
Brief Title: US Guided Erector Spinae Plane Block in Breast Cancer Surgery: Analgesia, Spread and Immunomodulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Mohamed Rabah Abdella, Principal investigator, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Medical Research Institute
Record Dates: First submitted 2020-11-24; First posted 2021-03-12 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Analgesia; Breast Cancer
Keywords: Erector spinae plane block; Ultrasound guided; Breast cancer surgery; Natural killer cells; Analgesia; spread
MeSH Terms: conditions — Agnosia; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ESPB Bubivacaine 0.25% (Experimental): 20 patients will receive US-guided deep ESPB block before induction of general anaesthesia using 20 ml bupivacaine 0.25 % and 5 ml of radiocontrast dye (Omnipaque) at the level of T4.
  Interventions: Procedure: Erector Spinae Plane Block with Bubivacaine
- ESPB Bubivacaine 0.125% (Active Comparator): 20 patients will receive US-guided deep ESPB block before induction of general anaesthesia using 40 ml bupivacaine 0.125 % and 5 ml of radiocontrast dye (Omnipaque) at the level of T4.
  Interventions: Procedure: Erector Spinae Plane Block with Bubivacaine
- No ESPB (Placebo Comparator): 20 patients will undergo standard general anaesthesia as a control group and postoperative analgesia with intravenous morphine patient controlled analgesia (PCA) and rescue analgesia if required.
  Interventions: Procedure: Standard General Anaesthesia

INTERVENTIONS:
Procedure: Erector Spinae Plane Block with Bubivacaine — Erector Spinae Plane Block with Bubivacaine 0.25% or 0.125% before breast cancer surgery
  Arms: ESPB Bubivacaine 0.125%; ESPB Bubivacaine 0.25%
Procedure: Standard General Anaesthesia — Standard General Anaesthesia without ESPB
  Arms: No ESPB

SUMMARY:
Prospective interventional study

DETAILED DESCRIPTION:
The aim of the present study is to evaluate the effect of US guided unilateral ESPB using different volumes of local anaesthetics on analgesic efficacy, dermatomal spread and immunomodulation in breast cancer surgery.

The primary outcome is the analgesic efficacy of the different local anaesthetic volumes of ESPB.

The secondary outcomes are the dermatomal dye spread and sensory coverage, immunomodulation and complications in breast cancer surgery.

Immunomodulation will be assessed by measuring Natural killer cells cytotoxicity.

ELIGIBILITY:
Inclusion Criteria:ASA physical status 1 or 2 scheduled for mastectomy under the effect of General Anaesthesia

-

Exclusion Criteria:

1. Patient refusal.
2. Allergy or contraindication to any of the studied medications or anaesthetic agents.
3. Chronic opioid analgesic use.
4. Pregnancy.
5. Morbid obesity (BMI ≥ 40 kg/m2).
6. Scoliosis or any vertebral anomalies or previous spinal surgeries.
7. Infection at the site of injection or any other contraindication for regional anaesthesia.
8. Duration of surgery more than 90 minutes.
9. Renal impairment.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2022-01-11 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
Analgesic efficacy of ESPB | Up to 24 postoperative hours
  Analgesic efficacy of Erector Spinae plabe block by measuring visual analogue scale which ranges from 0 to 10. 0 indicates no pain and 10 indicates maximum imaginable pain

SECONDARY OUTCOMES:
Spread of the injected dye in Erector Spinae plane | Patients will be imaged 15 minutes after the block and before induction of general anaesthesia and surgery.
  5 ml of radio-contrast dye will be injected in Erector Spinae plane with different dose of Bupivacaine at the level of 4th thoracic vertebra then spread of the dye will be assessed by CT scan (for example dye spread to first thoracic vertebra level cranially and 9th thoracic vertebra caudally).
  3 D reconstruction of the image will be done then Craniocaudal spread of the contrast and spread to Paravertebral space, epidural space or rami of the spinal nerves will be assessed and recorded.
Dermatomal sensory coverage of ESPB | Assessment will be done bilaterally every 3 minutes for 15 minutes after ESPB.
  will be assessed by hyposthesia to cold sensation. Field of sensory block from T1 to T6 will be assessed bilaterally every 3 minutes for 15 minutes after deep ESPB using a piece of cotton soaked in iced water. The adequacy of sensory block T1-T6 will be determined before induction of general anaesthesia.

OTHER OUTCOMES:
Immunomodulation of ESPB | Before ESPB and 24 hours after the block.
  Immunomodulation of ESPB by measuring Natural Killer cells cytotoxicity. Samples of 1 ml of patients' peripheral blood will be collected on EDTA for flow cytometry to enumerate for both cytotoxic lymphocyte populations (NK cells and cytotoxic t lymphocytes (Ctls)). CD 56 will be used as a marker for NK cells, while CD 8 will be used as a marker for Ctls.
  Cytotoxicity assay will be done by measuring the release of lactate dehydrogenase (LDH) from cells. Then ratio of LDH released specifically from NK cells will be correlated according to the results of flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Emad Eldin Abd El Monem Arida, Professor, Study Chair — University of Alexandria
Locations (1):
- Medical Research Institute, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: starting 6 months after publication

REFERENCES:
- [Derived] Abdella AMMR, Arida EEAEM, Megahed NA, El-Amrawy WZ, Mohamed WMA. Analgesia and spread of erector spinae plane block in breast cancer surgeries: a randomized controlled trial. BMC Anesthesiol. 2022 Oct 17;22(1):321. doi: 10.1186/s12871-022-01860-w. PMID 36253729

DOCUMENTS (1):
  • Study Protocol (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/63/NCT04796363/Prot_000.pdf